CLINICAL TRIAL: NCT05269264
Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema (LLL): Reliability, Concurrent Validity and Clinical Feasibility of Currently Applied Measurement Tools in Patients With LLL
Brief Title: Development of a Clinical Screening, Diagnostic and Evaluation Tool for Patients With Lower Limb Lymphedema: Aim 1
Acronym: EvaLymph-Leg1
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s66033-aim1
Record Dates: First submitted 2022-02-08; First posted 2022-03-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Lower Limb Lymphedema
Keywords: Lymphedema; Measurement; Clinical evaluation; Reliability; Concurrent validity; Clinical feasibility; Lower limb
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with unilateral or bilateral, primary or secundary lower limb lymphedema (LLL): patients with unilateral or bilateral, primary or secundary LLL who visit the center for lymphedema at UH Leuven
  Interventions: Diagnostic Test: Assessor A (first measurement): measurement methods and questionnaires for the assessment of LLL; Diagnostic Test: Assessor B: measurement methods and questionnaires for the assessment of LLL; Diagnostic Test: Assessor A (second measurement: measurement methods and questionnaires for the assessment of LLL
- healthy controls: age, BMI and gender matched to the patients with LLL
  Interventions: Diagnostic Test: Assessor A (first measurement): measurement methods and questionnaires for the assessment of LLL; Diagnostic Test: Assessor B: measurement methods and questionnaires for the assessment of LLL; Diagnostic Test: Assessor A (second measurement: measurement methods and questionnaires for the assessment of LLL
- subgroup (n=40): a subgroup of subjects (patients & healthy controls) will be evaluated again 2 weeks later
  Interventions: Diagnostic Test: Assessor A (first measurement): measurement methods and questionnaires for the assessment of LLL; Diagnostic Test: Assessor B: measurement methods and questionnaires for the assessment of LLL; Diagnostic Test: Assessor A (second measurement: measurement methods and questionnaires for the assessment of LLL; Diagnostic Test: Assessor A (2 weeks later): measurement methods and questionnaires for the assessment of LLL

INTERVENTIONS:
Diagnostic Test: Assessor A (first measurement): measurement methods and questionnaires for the assessment of LLL — pitting test at the level of the foot, leg and midline region; skinfold test at the level of the foot, leg and midline region; skin hardness test at the level of the foot, leg and midline region; measurement with MoistureMeterD at the level of the foot, leg and midline region; measurement with SkinFibroMeter at the level of the foot, leg and midline region; circumference measurements at the level of the leg and midline region; perometry at the level of the leg; water displacement measurement at the level of the foot; measurements with bio-impedance spectroscopy/analysis devices at the level of the lower limbs and a questionnaire regarding skin integrity (ICC compression questionnaire) that should be completed by the therapist and a self-reported disease-specific quality of life questionnaire (Lymph-ICF-LL) that is completed by the patient at the end of this evaluation
Diagnostic Test: Assessor B: measurement methods and questionnaires for the assessment of LLL — pitting test at the level of the foot, leg and midline region; skinfold test at the level of the foot, leg and midline region; skin hardness test at the level of the foot, leg and midline region; measurement with MoistureMeterD at the level of the foot, leg and midline region; measurement with SkinFibroMeter at the level of the foot, leg and midline region; circumference measurements at the level of the leg and midline region; perometry at the level of the leg; water displacement measurement at the level of the foot; measurements with bio-impedance spectroscopy/analysis devices at the level of the lower limbs and a questionnaire regarding skin integrity (ICC compression questionnaire) that should be completed by the therapist
Diagnostic Test: Assessor A (second measurement: measurement methods and questionnaires for the assessment of LLL — pitting test at the level of the foot, leg and midline region; skinfold test at the level of the foot, leg and midline region; skin hardness test at the level of the foot, leg and midline region; measurement with MoistureMeterD at the level of the foot, leg and midline region; measurement with SkinFibroMeter at the level of the foot, leg and midline region; circumference measurements at the level of the leg and midline region; perometry at the level of the leg; water displacement measurement at the level of the foot; measurements with bio-impedance spectroscopy/analysis devices at the level of the lower limbs and a questionnaire regarding skin integrity (ICC compression questionnaire) that should be completed by the therapist
Diagnostic Test: Assessor A (2 weeks later): measurement methods and questionnaires for the assessment of LLL — pitting test at the level of the foot, leg and midline region; skinfold test at the level of the foot, leg and midline region; skin hardness test at the level of the foot, leg and midline region; measurement with MoistureMeterD at the level of the foot, leg and midline region; measurement with SkinFibroMeter at the level of the foot, leg and midline region; circumference measurements at the level of the leg and midline region; perometry at the level of the leg; water displacement measurement at the level of the foot; measurements with bio-impedance spectroscopy/analysis devices at the level of the lower limbs and a questionnaire regarding skin integrity (ICC compression questionnaire) that should be completed by the therapist and a self-reported disease-specific quality of life questionnaire (Lymph-ICF-LL) that is completed by the patient at the end of this evaluation
  Groups: subgroup (n=40)

SUMMARY:
Of all of the different measurement methods that are currently available for use in clinical practice for assessing the same lymphedema characteristic (for example water displacement versus perimetry, both assessing swelling) or different lymphedema characteristics (for example water content in the skin versus hardness of the skin versus thickness of the skin), a clear overview about the reliability, concurrent validity (if applicable) and clinical feasibility is missing for the assessment of lower limb lymphedema (LLL).

The objective of this observational cross-sectional study is to investigate the (day-to-day) reliability and clinical feasibility of currently applied measurement tools in patients with LLL.

ELIGIBILITY:
Inclusion Criteria:

Patient group

* Unilateral or bilateral, primary or secondary Lower limb lymphedema (LLL)
* Objective diagnosis of lymphedema: ≥ 5% volume difference between both legs OR ≥ 2 minor/ 1 major criteria on lymphoscintigraphy OR presence of ICG dermal backflow
* Age ≥ 18 years
* Able to read, understand and speak Dutch

Healthy controls

- Age, gender & BMI-matched healthy controls

Exclusion Criteria:

* Pregnant participants
* Presence of chronic venous insufficiency C4, C5, C6; deep venous thrombosis; post-thrombotic syndrome
* Presence of skin infections of wounds at the level of the lower limbs at the moment of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with unilateral or bilateral, primary or secondary LLL will be recruited in the center for lymphedema in UH Leuven.
  The healthy controls will be age, gender & BMI matched subjects.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Within-session reliability of pitting test at the level of the foot, leg and midline region | baseline (within-session)
  intra and interrater reliability of pitting test at the level of the foot, leg and midline region;
  The grading of edema is determined by pit depth (measured visually) and recovery time from grade 0-3. The scale is used to rate the severity and the scores are as follows:
  - Grade 0: No clinical edema- Grade 1: Slight pitting (up to 2 mm depth) - Grade 2: Moderate pitting (2-5 mm) - Grade 3: Noticeably deep pit (>5 mm)
Within-session reliability of skinfold test at the level of the foot, leg and midline region | baseline (within-session)
  intra and interrater reliability of skinfold test at the level of the foot, leg and midline region Skin and subcutaneous tissue is lifted between thumb and index(and, if possible, compared to the contralateral side) Outcome:If skinfold is increased; yes(1), otherwise; no(0)
Within-session reliability of skin hardness test at the level of the foot, leg and midline region | baseline (within-session)
  intra and interrater reliability skin hardness test at the level of the foot, leg and midline region.
  Skin is palpated with thumb and index (and, if possible, compared to the contralateral side) Outcome: If skin is hardened; yes(1), otherwise; no(0)
Within-session reliability of measurement with MoistureMeterD at the level of the foot, leg and midline region | baseline (within-session)
  intra and interrater reliability of measurement with MoistureMeterD at the level of the foot, leg and midline region.
  This device can be applied to measure the percentage of water under the skin in terms of the Tissue Dielectric Constant value, making use of a probe with 300 MHz signal. Up to a depth of 2.5mm, this portable device allows measuring free and bounded water in the tissue through which the electromagnetic wave passes.
  Outcome: %PWC(% Percentage Water Content)
Within-session reliability of measurement with SkinFibroMeter at the level of the foot, leg and midline region | baseline (within-session)
  intra and interrater reliability of measurement with SkinFibroMeter at the level of the foot, leg and midline region.
  This device is a relatively recently developed device which consists of a 1-mm-long intender and records the resistance to 50 gram of pressure by using its reference plate and related built-in force sensors. Outcome: The resistance from the skin to deformation when an external force is applied, is expressed as a number in Newton (N) and represents the induration of the skin.
Within-session reliability of circumference measurements at the level of the leg and midline region | baseline (within-session)
  intra and interrater reliability of circumference measurements at the level of the leg and midline region; Outcome: in cm for each of the tapeline, but a total volume can be calculated (in ml) using a truncated cone formula
Within-session reliability of perometry at the level of the leg | baseline (within-session)
  intra and interrater reliability of perometry at the level of the leg; Optoelectronic volumetry (or perometry): a method that makes use of an optoelectronic infrared device to detect volume differences Outcome: in ml. The height of the measurement should be noted as well.
Within-session reliability of water displacement measurement at the level of the foot | baseline (within-session)
  intra and interrater reliability of water displacement measurement at the level of the foot
Within-session reliability of measurements with bio-impedance spectroscopy/analysis devices at the level of the lower limbs | baseline (within-session)
  intra and interrater reliability of measurements with bio-impedance spectroscopy/analysis devices at the level of the lower limbs
Within-session reliability of a questionnaire regarding skin integrity | baseline (within-session)
  intra and interrater reliability of a questionnaire regarding skin integrity (ICC compression questionnaire) that should be completed by the therapist The ICC-CQ is the first reliable and valid questionnaire evaluating different kinds of compression and the experience by patients with lymphedema or chronic venous disease.
Concurrent validity (only possible in case there are multiple measurement methods assessing the same lymphedema characteristic) of measurement methods for the assessment of LLL | baseline (within-session)
  the measurement methods assessing the same edema characteristic (for example: perometry and perimetry are two different methods that both evaluate lymphedema volume or swelling), will be correlated to each other
Clinical feasibility of measurement methods and questionnaires for the assessment of Lower lymb lymphoedema | baseline (within-session)
  Time efficiency will be examined for each method (timed), limitations regarding clinical feasibility will be listed and scored for each method (present or absent). Finally, an overall ranking regarding feasibility score will be determined based on the reliability (best -> worse reliability) and time-efficiency (fastest -> slowest measurement method).
Between-session reliability of pitting test at the level of the foot, leg and midline region | 2 weeks
  The grading of edema is determined by pit depth (measured visually) and recovery time from grade 0-3. The scale is used to rate the severity and the scores are as follows:
  - Grade 0: No clinical edema- Grade 1: Slight pitting (up to 2 mm depth) - Grade 2: Moderate pitting (2-5 mm) - Grade 3: Noticeably deep pit (>5 mm) A cohort of patients with LLL (n= ±40) and healthy volunteers (±40) will be scheduled for a second visit, 2 weeks later for the same clinical evaluation (as at baseline), with only 1 assessor.
Between-session reliability of skinfold test at the level of the foot, leg and midline region | 2 weeks
  Skin and subcutaneous tissue is lifted between thumb and index(and, if possible, compared to the contralateral side) Outcome:If skinfold is increased; yes(1), otherwise; no(0)
  A subgroup of patients with LLL (n= ±40) and healthy volunteers (±40) will be scheduled for a second visit, 2 weeks later for the same clinical evaluation (as at baseline), with only 1 assessor.
Between-session reliability of skin hardness test at the level of the foot, leg and midline region | 2 weeks
  Skin is palpated with thumb and index (and, if possible, compared to the contralateral side) Outcome: If skin is hardened; yes(1), otherwise; no(0)
  A subgroup of patients with LLL (n= ±40) and healthy volunteers (±40) will be scheduled for a second visit, 2 weeks later for the same clinical evaluation (as at baseline), with only 1 assessor.
Between-session reliability of measurement with MoistureMeterD at the level of the foot, leg and midline region | 2 weeks
  This device can be applied to measure the percentage of water under the skin in terms of the Tissue Dielectric Constant value, making use of a probe with 300 MHz signal. Up to a depth of 2.5mm, this portable device allows measuring free and bounded water in the tissue through which the electromagnetic wave passes.
  Outcome: %PWC(% Percentage Water Content)
  A subgroup of patients with LLL (n= ±40) and healthy volunteers (±40) will be scheduled for a second visit, 2 weeks later for the same clinical evaluation (as at baseline), with only 1 assessor.
Between-session reliability of measurement with SkinFibroMeter at the level of the foot, leg and midline region | 2 weeks
  This device is a relatively recently developed device which consists of a 1-mm-long intender and records the resistance to 50 gram of pressure by using its reference plate and related built-in force sensors. Outcome: The resistance from the skin to deformation when an external force is applied, is expressed as a number in Newton (N) and represents the induration of the skin.
  A subgroup of patients with LLL (n= ±40) and healthy volunteers (±40) will be scheduled for a second visit, 2 weeks later for the same clinical evaluation (as at baseline), with only 1 assessor.
Between-session reliability of circumference measurements at the level of the leg and midline region | 2 weeks
  Circumference measurements (cm) with perimeter.
  A subgroup of patients with LLL (n= ±40) and healthy volunteers (±40) will be scheduled for a second visit, 2 weeks later for the same clinical evaluation (as at baseline), with only 1 assessor.
Between-session reliability of perometry at the level of the leg | 2 weeks
  Optoelectronic volumetry (or perometry): a method that makes use of an optoelectronic infrared device to detect volume differences Outcome: in ml. The height of the measurement should be noted as well.
  A subgroup of patients with LLL (n= ±40) and healthy volunteers (±40) will be scheduled for a second visit, 2 weeks later for the same clinical evaluation (as at baseline), with only 1 assessor.
Between-session reliability of water displacement measurement at the level of the foot | 2 weeks
  'Gold standard' in which the limb is immersed into a water tank and the weight of the limb is being weighted.
  A subgroup of patients with LLL (n= ±40) and healthy volunteers (±40) will be scheduled for a second visit, 2 weeks later for the same clinical evaluation (as at baseline), with only 1 assessor.
Between-session reliability of measurements with bio-impedance spectroscopy/analysis devices at the level of the lower limbs | 2 weeks
  Bio-impedance spectroscopy assesses the resistance (or impedance) to the flow of an electrical current that is primarily conducted by body fluid.
  A subgroup of patients with LLL (n= ±40) and healthy volunteers (±40) will be scheduled for a second visit, 2 weeks later for the same clinical evaluation (as at baseline), with only 1 assessor.
Between-session reliability of a questionnaire regarding skin integrity | 2 weeks
  Between-session reliability of a questionnaire regarding skin integrity: ICC compression questionnaire that should be completed by the therapist The ICC-CQ is the first reliable and valid questionnaire evaluating different kinds of compression and the experience by patients with lymphedema or chronic venous disease
Between-session reliability of a self-reported disease-specific quality of life questionnaire (Lymph-ICF-LL) | 2 weeks
  The Lymph-ICF-LL is a descriptive, evaluative tool containing 28 questions about impairments in function, activity limitations, and participation restrictions in patients with lower limb lymphedema. The questionnaire has 5 domains: physical function, mental function, general tasks/household activities, mobility activities, and life domains/social life.

CONTACTS AND LOCATIONS:
Overall Officials: Tessa De Vrieze, Dr., Principal Investigator — KU Leuven
Locations (1):
- University Hospitals of Leuven, center for lymphedema, Leuven, Belgium